CLINICAL TRIAL: NCT06612359
Title: Impact of the BOOST GAIT Program on Gait Recovery and Functional Mobility After Stroke - a Pilot Study Impact Van Het BOOST GAIT Programma Op Het Herstel Van Het Gangbeeld En Functionele Mobiliteit Na Een Beroerte - Een Pilootstudie
Brief Title: Impact of the BOOST GAIT Program on Gait Recovery and Functional Mobility After Stroke
Acronym: BOOST GAIT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Peter Feys, Professor Rehabilitation Sciences, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/029 - BOOST GAIT pilot; B2432024000003 (Other: Belgian registration number)
Record Dates: First submitted 2024-08-30; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Stroke with Hemiparesis; Stroke
Keywords: Recovery; Gait; Physical exercise; Pilot study; Stroke; Hemiparesis; Walking
MeSH Terms: conditions — Stroke; Motor Activity; Paresis

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BOOST GAIT (Experimental): Participants recruited for this pilot study will undergo the BOOST GAIT program in addition to their usual inpatient rehabilitation care.
  Interventions: Behavioral: BOOST GAIT Program

INTERVENTIONS:
Behavioral: BOOST GAIT Program — In addition to usual care, participants will undergo additional therapy over a four-week period, with sessions occurring five times per week for one hour. The BOOST GAIT sessions will be conducted as group-based therapy with four patients and two physiotherapists present to oversee the performance of mobility-specific exercises, including sit-to-stand transfers, standing and stepping, and eventually walking.

SUMMARY:
The overarching goal is to determine if the BOOST GAIT program can improve functional mobility in patients with stroke who are undergoing inpatient rehabilitation and have some walking function, through the application of augmented therapeutic exercises designed to achieve a normative gait pattern. The evaluation will be conducted using a combination of clinical scales and objective motion sensors that map walking quality and performance during activities of daily living, such as rising from a chair and standing.

It is acknowledged that this single-group pilot study, which aims to include 12 participants, is insufficiently powered to address the primary objective. A larger parallel-design study is required to definitively address this issue. To help design a larger study, the current objectives are: first, to have realistic expectations regarding recruitment and dropout rates; second, to identify potential barriers to therapy adherence and data collection that may impede the success of a larger study; third, assess the test-retest reliability of sensor-based motion capture of movement quality during walking and related tasks in hemiparetic stroke patients. For the latter objective, the sensor measurements at the end of the intervention will be repeated on two consecutive days.

In addition to their usual care, participants will undergo additional therapy over a four-week period, with sessions occurring five times per week for one hour as part of the BOOST GAIT program. The BOOST GAIT sessions will be conducted as group-based therapy with four patients and two physiotherapists present to oversee the performance of mobility-specific exercises, including sit-to-stand transfers, standing and stepping, and eventually walking. The rationale for this approach is that the combined effects of augmenting the amount of therapeutic exercises and specifically targeting motor control of the paretic leg will facilitate symmetry during tasks, which in turn will have carry-over effects on safe performance of walking and other mobility tasks.

ELIGIBILITY:
Inclusion Criteria:

* A first-ever unilateral stroke, infarction or bleeding
* Undergoing inpatient rehabilitation in the Jessa hospital, Herk-de-Stad
* Less than 3 months after stroke onset at the moment of inclusion
* 18 years of older
* Berg Balance Scale score 24 or higher (out of 56) at moment of inclusion
* Timed Up-and-Go score 14 s or higher at moment of inclusion
* Functional Ambulation Category 3 or higher at moment of inclusion
* Understanding the goals and procedures of this study and giving informed consent

Exclusion Criteria:

* Significant cognitive and/or speech impairments that markedly affect the comprehension and execution of instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-selected Gait Speed (m/s) | At inclusion and the end of the intervention at 4 weeks.
  The 10-meter walk test (10m-WT) is used as a performance measure to assess gait speed in meters per second over a short distance. We follow a standardized protocol with 3 immediate test-retest repetitions while the participant is instructed to walk safely at a comfortable pace.

SECONDARY OUTCOMES:
Fugl-Meyer assessment - motor subscale for the Lower Extremity (FM-LE) [0-34] | At inclusion and the end of the intervention at 4 weeks.
  The FM-LE is a stroke-specific impairment measure that assesses the ability to produce voluntary movement control outside of synergistic patterns. A score of 0 indicates a completely flaccid, paralyzed limb, whereas a score of 34 reflects full motor function with synergy-independent movement. A higher score therefore reflects a better outcome.
Motricity Index - subscale for the Lower Extremity (MI-LE) [0-100] | At inclusion and the end of the intervention at 4 weeks.
  The MI-LE is an impairment measure that assesses the ability to produce maximum muscle force in the direction of hip flexion, knee extension, and ankle dorsiflexion. Each item is with a score of 0 indicating a paralyzed limb and a score of 33 reflecting normal strength against manual resistance. The maximum score of 99 is set to 100 to give an index score in % of the degree of strength impairment. A higher score therefore reflects a better outcome.
Berg Balance Scale (BBS) [0-56] | At inclusion and the end of the intervention at 4 weeks.
  The BBS is used to rate the ability to safely balance during 14 predetermined tasks. Each task is evaluated on a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. A higher score therefore reflects a better outcome.
Functional Ambulation Category (FAC) [0-5] | At inclusion and the end of the intervention at 4 weeks.
  The FAC is a 6-point scale determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. A score of 0 means total disability, whereas a maximum score of 5 mean full independent walking over uneven terrains. A higher score therefore reflects a better outcome.
Smoothness during a sit-to-stand transfer | At inclusion and the end of the intervention at 4 weeks.
  A wearable sensor system (APDM, Opal sensors) will be used to measure quality indicators of smoothness of a sit-to-stand transition. For this purpose, sensors will be attached to the body while recording kinematic data during standing-up from a chair of standardized height without using the arms. The participant is instructed to do this as fast as possible. Shorter and smoother motion mean a better outcome.
Postural sway during quiet standing | At inclusion and the end of the intervention at 4 weeks.
  A wearable sensor system (APDM, Opal sensors) will be used to measure the amount of body sway during a quiet stance task. For this purpose, sensors will be attached to the body while kinematic data will be measured during standing with the feet placed at shoulder width. The participant is instructed to remain as still as possible. Reduced levels of sway mean a better outcome.
Spatio-temporal parameters of the gait pattern during self-selected walking over a short distance | At inclusion and the end of the intervention at 4 weeks.
  A wearable sensor system (APDM, Opal sensors) will be used to measure spatio-temporal aspects of the gait pattern, with particular interest in estimates of interlimb symmetry, over a short distance. For this purpose, the sensors are attached to the body to record the motion kinematics during a straight, unobstructed walk. The participant is instructed to walk at comfortable pace for 30 seconds. Longer, faster and more consistent steps (ie, less variability), with more symmetry between the legs, mean a better outcome.
Spatio-temporal parameters of the gait pattern during fastest walking over a longer distance | At inclusion and the end of the intervention at 4 weeks.
  A wearable sensor system (APDM, Opal sensors) will be used to measure spatio-temporal aspects of the gait pattern, with particular interest in estimates of interlimb symmetry, over a longer distance. For this purpose, the sensors are attached to the body to record the motion kinematics during a straight, unobstructed walk. The participant is instructed to walk as fast as possible, continuously for 3 minutes. Longer, faster, more consistent and symmetric steps, without decrement over the 3-min period as reflections of fatigue, mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, Professor, Principal Investigator — Hasselt University, REVAL Rehabilitation Research center; Maaiken Vander Plaetse, MD, Principal Investigator — FRAME, Jessa Hospital
Locations (1):
- FRAME by Jessa Ziekenhuis, Herk-de-Stad, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No